CLINICAL TRIAL: NCT05922592
Title: Balloon Technique Versus Densah Bur in Crestal Sinus Lift Operation With Simultaneous Implant Placement. A Prospective Study
Brief Title: Different Techniques of Crestal Sinus Lift
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed mahmoud alajami, postgraduate student at oral an maxillofacial surgery department, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A08030123
Record Dates: First submitted 2023-06-19; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Crestal Sinus Lift

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The sinus membrane will be elevated by using balloon technique with simultaneous Implant placement. (Experimental)
  Interventions: Procedure: crestal sinus lift using ballon technique
- The sinus membrane will be elevated by using Densah burs with simultaneous Implant placement (Experimental)
  Interventions: Procedure: crestal sinus lift using densah burs

INTERVENTIONS:
Procedure: crestal sinus lift using ballon technique — The sinus membrane will be elevated by using balloon technique with simultaneous Implant placement.
  Arms: The sinus membrane will be elevated by using balloon technique with simultaneous Implant placement.
Procedure: crestal sinus lift using densah burs — The sinus membrane will be elevated by using Densah burs with simultaneous Implant placement
  Arms: The sinus membrane will be elevated by using Densah burs with simultaneous Implant placement

SUMMARY:
Sixteen patients will be selected from those attending the outpatient clinic of the Oral & Maxillofacial Surgery Department, Faculty of Dentistry, Mansoura University with age range from 20-50 years seeking implantation of their lost posterior maxillary teeth, [premolar and molars] with limited bone height below the floor of the maxillary sinus, secondary to sinus pneumatization.

Group I (N = 8): The sinus membrane will be elevated by using balloon technique with simultaneous Implant placement.

Group II (N = 8): The sinus membrane will be elevated by using Densah burs with simultaneous Implant placement.

ELIGIBILITY:
Inclusion Criteria:

* Patent ostium of maxillary sinus.
* Patient with missing one or more posterior maxillary teeth.
* A ridge height at the site of implantation of 4-7 mm.
* A ridge width at the site of implantation of 6 mm.
* Good oral hygiene.
* Patients in the age frame between 20 years and 50 years old.
* No gender preface in selection of the patients.
* Acceptable inter-arch space for the future prosthesis.

Exclusion Criteria:

* Any pathological condition at the site of surgery.
* Patients with systemic diseases that contra-indicate the surgical procedure such as uncontrolled diabetes mellitus, bleeding disorders, serious osseous disorders, and mental disorders.
* Heavy smoking and alcoholism.
* Parafunctional habits such as bruxism and clenching.
* Signs of acute infection or pus discharge
* Disturbed occlusion.
* Maxillary sinus inflammation.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Height gain | 6 months
  Bone height after the surgery measured on CBCT 6-months postoperative _ Residual bone height at implant placement

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Mahmoud, Al Mansurah, Egypt

REFERENCES:
- [Derived] Alajami MM, Elsheikh HA, Abo El-Farag SA, Mansour NA. Antral membrane balloon technique versus Densah bur in crestal sinus lift with simultaneous implant placement: a randomized clinical trial. BMC Oral Health. 2024 Aug 8;24(1):916. doi: 10.1186/s12903-024-04609-8. PMID 39118095